CLINICAL TRIAL: NCT04164030
Title: Merging Yoga, Occupational Therapy and Education in Diabetes Management
Brief Title: Education and Exercise Program for Adults With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado State University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140898
Record Dates: First submitted 2019-09-16; First posted 2019-11-15 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
Keywords: low income adults; feasibility pilot study; occupational therapy; nutrition education; yoga
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status; Nutrition Assessment; Occupational Therapy; Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education Control (Active Comparator): An evidence-based nutrition program entitled Eating Smart Being Active. Delivered in a group: Meets weekly for 2 hours for 9 weeks.
  Interventions: Behavioral: Education and Exercise Program for Adults with Type 2 Diabetes
- Nutrition Education +OT+Yoga (Experimental): 9 week group that meets twice a week for two hours each. Group occupational therapy and group yoga will be added to the nutrition program.
  Interventions: Behavioral: Nutrition Education plus Occupational Therapy plus Yoga

INTERVENTIONS:
Behavioral: Education and Exercise Program for Adults with Type 2 Diabetes — Eating Smart and Being Active program
  Arms: Nutrition Education Control
Behavioral: Nutrition Education plus Occupational Therapy plus Yoga — multimodal interdisciplinary approach
  Arms: Nutrition Education +OT+Yoga

SUMMARY:
The purpose of this two phase study is to: 1) develop and 2) assess a program titled: Merging Yoga, Occupational Therapy and Nutrition Education (MY-OT-Ed) designed for low income adults with Type 2 Diabetes. Half of the participants will participate in the Nutrition Education, and the other half of the participants will participate in Nutrition Education plus Occupational Therapy group and group yoga.

DETAILED DESCRIPTION:
Merging Yoga, Occupational Therapy and Nutrition Education (MY-OT-Ed) is an interdisciplinary program designed to help low income adults with Type 2 Diabetes engage fully in life while learning to manage their diabetes. The aim is to empower individuals to embed diabetes self-management into everyday activities and routines while upholding quality of life. Currently Extension Services bring nutrition education to the under-served population in the local communities through the Expanded Food and Nutrition Education Program (EFNEP). Colorado EFNEP uses the evidence-based, healthy eating and active living curriculum, Eating Smart • Being Active (ESBA), with adult participants. While EFNEP may be helpful in the management of some aspects of diabetes care, it is not designed to address the established self-care behaviors and routines essential for effective diabetes self management. Therefore, it is critical to merge nutrition education programs such as EFNEP with other established interventions to best meet the needs of the individual with diabetes. Likewise, yoga is an effective form of physical activity to manage some aspects of diabetes care and outcomes. However, yoga is also not enough to address all of the needs of the individual. Furthermore, evidence for the success of occupational therapy's role in diabetes self-management is growing as a way to manage some aspects of the complexity of diabetes care or routines in everyday life. Our aim in this study is to follow best practice and create and evaluate an interdisciplinary approach to type 2 diabetes self-management by merging together yoga, occupational therapy and nutritional education to improve diabetes related outcomes in our population.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak English and answer questions/communicate
* Self-report diagnosis of Type 2 Diabetes
* Self-report of children living at home
* Self-report of low socioeconomic status or use of food assistance programs

Exclusion Criteria:

* pregnant or anticipation of becoming pregnant in the next 6 months
* completion of Type 2 Diabetes self-management or participation in occupational therapy with an emphasis on managing diabetes or other chronic condition in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in habits measured using the Self-Report Habit Index | Pre assessment, post assessment following 9 week session and 6-8 weeks follow-up
  The Self-Report Habit Index contains 12 items that measures habit strength, including automaticity, repeated character of the behavior and the sense of identity the behavior reflects. A 5 point likert scale (ranging from strongly agree (4), to strongly disagree (0) ) is used to score each item. The Self-Report Habit Index yields a total score by summing all of the items together. The total score ranges from 0 - 48, with a higher score representing a stronger habit.
Change in diabetes distress measured using the Diabetes Distress Scale | Pre assessment, post assessment following 9 week session and 6-8 weeks follow-up
  The Diabetes Distress Scale contains 17 items, which assess causes of burden and worries related to managing a chronic disease as diabetes. A 6 point likert scale (1 = no problem; 6 = severe problem) is used to score each item. The Diabetes Distress Scale yields a total score and 4 sub scale scores, including emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. The total score and sub scale scores are calculated by summing the responses of the number of items and dividing by the number of items. There are five items for emotional burden, 4 items for physician-related distress, 5 items for regimen-related distress, and 3 items for interpersonal distress. Therefore, the total and sub-scores are each reported as a mean item score, ranging from 1-6, with a higher score representing greater distress reported.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Atler, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States